CLINICAL TRIAL: NCT03566485
Title: BRE 17107: A Phase Ib/II Trial of Atezolizumab (an Anti-PD-L1 Monoclonal Antibody) With Cobimetinib (a MEK1/2 Inhibitor) or Idasanutlin (an MDM2 Antagonist) in Metastatic ER+ Breast Cancer
Brief Title: Atezolizumab and Cobimetinib or Idasanutlin in Participants With Stage IV or Unresectable Recurrent Estrogen Receptor Positive Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual/Loss of funding
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Stand Up To Cancer (Other)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 17107; NCI-2018-01159 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Estrogen Receptor-positive; HER2/Neu Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; cobimetinib; RG7388

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 2 (atezolizumab, cobimetinib) (Experimental): Participants with TP53 gene mutation receive atezolizumab IV over 60 minutes starting with day 15 of course 1 and then on days 1 and 15 of subsequent courses, and cobimetinib PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib
- Phase 1b - Atezolizumab 840mg IV + Idasanutlin 100mg PO (Experimental)
  Interventions: Drug: Atezolizumab; Drug: Idasanutlin

INTERVENTIONS:
Drug: Atezolizumab — Given by IV
Drug: Cobimetinib — Given by mouth
  Arms: Phase 2 (atezolizumab, cobimetinib)
Drug: Idasanutlin — Given by mouth
  Arms: Phase 1b - Atezolizumab 840mg IV + Idasanutlin 100mg PO

SUMMARY:
This phase I/II trial studies the side effects and best dose of idasanutlin when given together with atezolizumab, and to see how well atezolizumab and cobimetinib or idasanutlin work in treating participants with stage IV estrogen-receptor positive (ER+) breast cancer, or ER+ breast cancer that has come back (recurrent) and cannot be removed by surgery (unresectable). Monoclonal antibodies, such as atezolizumab, may interfere with the ability of tumor cells to grow and spread. Cobimetinib and idasanutlin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving atezolizumab with cobimetinib or atezolizumab with idasanutlin may work better in treating participants with estrogen-receptor positive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of atezolizumab and idasanutlin in patients with estrogen receptor positive (ER+) metastatic breast cancer (mBC) (Phase I).

II. To determine the anti-tumor effect of atezolizumab and cobimetinib or idasanutlin in patients with ER+ mBC (Phase II).

SECONDARY OBJECTIVES:

I. To determine the anti-tumor duration of effect of atezolizumab and cobimetinib or idasanutlin in patients with ER+ mBC (Phase II).

II. To determine the safety and tolerability of atezolizumab and cobimetinib or idasanutlin in patients with ER+ mBC (Phase II).

EXPLORATORY OBJECTIVES:

I. To evaluate if CD8+ T cells are enhanced in the tumor with either MEK or MDM2 inhibition (Phase II).

II. To evaluate if MHC-I/II and/or PD-L1 expression is enhanced with MEK inhibition (Phase II).

III. To evaluate if T cell chemotractants (CCL5, CXCL9,10,11,13) are upregulated upon MDM2 antagonism (Phase II).

IV. To determine if baseline or changes in PDL1 expression, MHC expression, presence of tumor infiltrating lymphocytes, neoantigen expression/ mutation burden (using ribonucleic acid [RNA]-and whole exome sequencing), CCL5, CXCL9, CXCL10, CXCL11, and CXCL13 correlate with clinical outcome (Phase II).

V. To determine if immunological activity of MEK inhibition can be tracked noninvasively using Zr^89-atezolizumab (Phase II).

OUTLINE: This is a phase 1, dose-escalation study of idasanutlin followed by a phase II study. Participants are assigned to 1 of 2 arms.

ARM I: Participants with TP53 gene mutation receive atezolizumab intravenously (IV) over 60 minutes starting with day 15 of course 1 and then on days 1 and 15 of subsequent courses, and cobimetinib orally (PO) daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Participants without TP53 gene mutation receive atezolizumab IV over 60 minutes starting with day 15 of course 1 and then on days 1 and 15 of subsequent courses, and idasanutlin PO daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed for 28 days.

ELIGIBILITY:
* Signed and dated written informed consent.
* Subjects ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Clinical stage IV invasive mammary carcinoma or unresectable locoregional recurrence of invasive mammary carcinoma that is:

  * ER/PR-positive (> 1% cells) by IHC and HER2 negative per ASCO guidelines (by IHC or FISH)
  * Previously exposed to an aromatase inhibitor (AI) or a selective estrogen-receptor modulator/ downregulator (SERM; SERD) + a CDK4/6 inhibitor
  * Appropriate candidates for chemotherapy
  * Amenable to biopsy at the time of study entry
* Adequate organ function including:

  * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
  * Platelets ≥ 100 × 109/L
  * Hemoglobin ≥ 9/g/dL (may have been transfused)
  * Total serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 2.5 × ULN (or ≤ 5 × ULN if liver metastases are present)
  * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 50 mL/min as calculated using the Cockcroft-Gault (CG) equation
  * Thyroid Stimulating Hormone (TSH) ≤ 1 x ULN
  * Amylase ≤ 1 x ULN
  * Lipase ≤ 1 x ULN
  * CPK ≤ 1.5 x ULN
  * LVEF (echo) ≥ LLN (Cobi arm only)
* Female patients of childbearing potential must agree to use at least two methods of acceptable contraception with a failure rate of < 1% per year from 15 days prior to first trial treatment administration until at least 5 months after study participant's final dose of study drugs. See appendix C for details.

Note: Females of childbearing potential are defined as those who are not surgically sterile or post-menopausal (i.e. patient has not had a bilateral tubal ligation, a bilateral oophorectomy, or a complete hysterectomy; or has not been amenorrheic for 12 months without an alternative medical cause). Post-menopausal status in females under 55 years of age should be confirmed with a serum follicle-stimulating hormone (FSH) level within laboratory reference range for postmenopausal women.

* Patients unable to read/write in English are eligible to participate in the overall study but will not participate in the Patient-Reported Outcome questionnaires throughout the trial
* Re-enrollment of a subject that has discontinued the study as a pre-treatment screen failure (i.e. a consented patient who did not receive study drugs) is permitted. If re-enrolled, the subject must be re-consented. Only the screening procedures performed outside of protocol-specified timing must be repeated.

Exclusion Criteria:

* Prior therapy with anti-PD-L1 and anti-PD1 antibodies, MEK inhibitors or MDM2 antagonists.
* No more than 3 lines of chemotherapy in the metastatic setting
* No concurrent anticancer therapy. Required washout from prior therapy:

  * Endocrine therapy: no required wash-out
  * Chemotherapy: 14 days
  * Major surgery: 14 days (provided wound healing is adequate)
  * Radiation: 7 days
  * Investigational/Biologic Therapy (half -life ≤ 40 hours): 14 days
  * Investigational/Biologic Therapy (half -life > 40 hours): 28 days
  * Use of corticosteroids or immunosuppressive medication is exclusionary, except the following in the absence of active autoimmune disease:

    * Subjects are permitted the use of corticosteroids with minimal systemic absorption (e.g. topical, ocular, intra-articular, intranasal, and inhaled);
    * Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent are permitted;
    * Adrenal replacement steroid doses including doses > 10 mg daily prednisone are permitted;
    * A brief (less than 3 weeks) course of corticosteroids for prophylaxis (e.g. CT scan premedication against contrast dye allergy) or for treatment of non-autoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by a contact allergen) is permitted.
* Previous malignant disease other than breast cancer within the last 5 years, with the exception of basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, or low-risk cancers considered curatively treated (i.e. complete remission achieved at least 2 years prior to first dose of study drugs AND additional therapy not required while receiving study treatment).
* All subjects with brain metastases, except those meeting the following criteria:

  * Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrollment
  * No history of intracranial or spinal cord hemorrhage
  * No evidence of interim CNS disease progression
  * Metastasis to the midbrain, pons, and medulla
  * No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable.
  * Subjects must be either off steroids or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent)
* Receipt of any organ transplantation including allogeneic stem-cell transplantation.
* Significant acute or chronic infections including, among others:

  * Known history of testing positive for human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS).
  * Active tuberculosis
  * Positive test for hepatitis B virus (HBV) surface antigen (and/or core antibody) and/or confirmatory hepatitis C virus (HCV) RNA (if anti-HCV antibody tested positive).
* Active autoimmune disease with reasonable possibility of clinically significant deterioration when receiving an immunostimulatory agent:

  * Subjects with Type 1 diabetes mellitus, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
  * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day.
  * Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable.
* Interstitial lung disease that is symptomatic or which may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Uncontrolled asthma [defined as having 3 or more of the following features of partially controlled asthma within 28 days prior to starting study treatment: Daytime symptoms more than twice per week, any limitation of activities, any nocturnal symptoms/awaking, need for reliever/rescue inhaler more than twice per week, or known lung function (PEF or FEV1) without administration of a bronchodilator that is < 80% predicted or personal best (if known)].
* Current symptomatic congestive heart failure (New York Heart Association > class II), unstable cardiac arrhythmia requiring therapy (e.g. medication or pacemaker), unstable angina (e.g. new, worsening or persistent chest discomfort), or uncontrolled hypertension (systolic > 160 mmHg or diastolic > 100mmHg). Or any of the following occurring within 6 months (180 days) prior to first dose of study drugs: Myocardial infarction, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack. (Use of antihypertensive medication to control blood pressure is allowed.)
* Concurrent treatment with a non-permitted drug (refer to prohibited medication list) as well as foods or supplements that are strong or moderate CYP3A4 enzyme inducers or inhibitors. Any of the above has to be discontinued at least 7 days prior to Cycle 1/ Day 1 of study treatment.
* Requirement of anticoagulant therapy with oral vitamin K antagonists such as Coumadin (warfarin). Low-dose anticoagulants for the maintenance of patency in a central venous access device or the prevention of deep vein thrombosis or pulmonary embolism is allowed. Therapeutic use of low molecular weight heparin is allowed provided patients are safely able to interrupt it prior to biopsy procedures.
* Persisting toxicity related to prior therapy that has not reduced to Grade 1 [National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 5.0]; however, alopecia and sensory neuropathy Grade ≤ 2 are acceptable and Grade ≤ 2 non-hematological toxicities well controlled with medical management are allowed (for example: hypomagnesemia well controlled on magnesium replacement).
* Known severe (Grade ≥ 3 NCI-CTCAE) hypersensitivity reactions to monoclonal antibodies, or history of anaphylaxis.
* Vaccination within 28 days of the first dose of study drugs and while on trial is prohibited, except for administration of inactivated vaccines (for example, inactivated influenza vaccine).
* Pregnant or breastfeeding females.
* Known current alcohol or drug abuse
* Prisoners or subjects who are involuntarily incarcerated.
* Known psychiatric condition, social circumstance, or other medical condition reasonably judged by the patient's study physician to unacceptably increase the risk of study participation; or to prohibit the understanding or rendering of informed consent or anticipated compliance with scheduled visits, treatment schedule, laboratory tests and other study requirements.
* Known risk factors for ocular toxicity, consisting of any of the following (Cobi arm only):

  * presence of serous retinopathy within 6 months of protocol enrollment
  * presence of retinal vein occlusion (RVO) within 6 months of protocol enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to this study from July 2018 to November 2019 at Vanderbilt-Ingram Cancer Center in Nashville, TN. This study stopped early due to low accrual.
Pre-assignment Details: Twelve participants were enrolled onto this study.
Groups:
- Phase 1b - (Atezolizumab, Idasanutlin): Atezolizumab: Given by IV
  Idasanutlin: Given by mouth
Period: Overall Study
Arm/Group | Phase 2 (Atezolizumab, Cobimetinib) | Phase 1b - (Atezolizumab, Idasanutlin)
Started | 5 | 7 (Dose level 1 (Idasanutlin 100mg PO))
Completed | 0 | 0
Not Completed | 5 | 7
Not completed — Disease progression | 5 | 4
Not completed — Clinical progression | 0 | 1
Not completed — Toxicity | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 2 (Atezolizumab, Cobimetinib) | Phase 1b - (Atezolizumab, Idasanutlin) | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT) (Phase I)
Description: Assessment of DLT for the patients in the atezolizumab and idasanutiln arm of the study
Time Frame: At 28 days
Population: patients in the atezolizumab and idasanutiln arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b - (Atezolizumab, Idasanutlin)
Number analyzed (Participants) | 7
Participants | 1

2. Primary Outcome: Maximum Tolerated Dose (Phase I)
Description: Assessment of MTD for the atezolizumab and idasanutiln combination arm of the study
Time Frame: At 28 days
Population: Patients in the atezolizumab and idasanutiln combination arm of the study. Dosage used: Atezolizumab 840mg IV + Idasanutlin 100mg PO
Measure: Number; unit: mg
Arm/Group | Phase 1b - (Atezolizumab, Idasanutlin)
Number analyzed (Participants) | 7
mg | NA — Not enough patients were put on the Idasa + Atezo arm; therefore, unable to determine MTD. Dosage used: Atezolizumab 840mg IV + Idasanutlin 100mg PO.

3. Primary Outcome: Recommended Phase II Dose (Phase I)
Description: Assessment of recommended phase II dose for the atezolizumab and idasanutiln combination arm of the study
Time Frame: At 28 days
Population: Patients on the atezolizumab and idasanutiln combination arm of the study. Dosage used: Atezolizumab 840mg IV + Idasanutlin 100mg PO.
Measure: Number; unit: mg
Arm/Group | Phase 1b - (Atezolizumab, Idasanutlin)
Number analyzed (Participants) | 7
mg | NA — Not enough patients were put on the Idasa + Atezo arm; therefore, unable to determine MTD and recommend dose for phase II. Dosage used: Atezolizumab 840mg IV + Idasanutlin 100mg PO. For phase II, no patients were assigned to this arm.

4. Primary Outcome: Overall Response Rate (ORR; by Response Evaluation Criteria in Solid Tumors [RECIST]1.1) (Phase II)
Description: Assessment of clinical impact (anti-tumor effect) of the combination of atezolizumab and cobimetinib or idasanutiln in patients with metastatic ER
  + breast cancer by measure the rate (%) of complete and partial responses seen in patients with measurable disease. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 28 days after completion of study treatment, for a total of 2 years
Population: Patients on Phase 2 Arm 1 (TP53-mut) - Atezolizumab 840mg IV + Cobimetinib 60mg PO
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 5
percentage of participants | NA [NA to NA] — Among the 5 participants, two patients had only baseline measurements, one patient had only follow up measurement, and one patient did not have any measurements. Only one patient had progressive disease after baseline measurement. Therefore, not enough number of patients for calculating this outcome.

5. Secondary Outcome: Clinical Benefit Rate (CBR) (Phase II)
Description: Assessment of clinical impact (anti-tumor effect) of the combination of atezolizumab and cobimetinib or idasanutiln in patients with metastatic ER
  + breast cancer by measure the rate (%) of complete and partial responses + stability of disease at 6 months seen in patients with measurable disease. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: At 6 months
Population: patients on Phase 2 Arm 1 (TP53-mut) - Atezolizumab 840mg IV + Cobimetinib 60mg PO
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 5
percentage of participants | NA [NA to NA] — Among 5 participants, two patients had only baseline measurements, one patient had only follow up measurement, and one patient did not have any measurements. Only one patient had progressive disease after baseline measurement. Therefore, not enough number of patients for calculating this outcome.

6. Secondary Outcome: Immune Related Response Criteria (irRC) (Phase II)
Description: Assessment of clinical impact (anti-tumor effect) of the combination of atezolizumab and cobimetinib or idasanutiln in patients with metastatic ER
  + breast cancer by measure the rate (%) of immune-related complete and partial responses seen in patients with measurable disease
Time Frame: Up to 28 days after completion of study treatment, for a total of 2 years
Population: An insufficient number of participants exhibited response for analysis.
Arm/Group | Phase 2 (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 0

7. Secondary Outcome: Progression-free Survival (PFS) (Phase II) in Days
Description: Assessment of clinical impact (anti-tumor effect) of the combination of atezolizumab and cobimetinib or idasanutiln in patients with metastatic ER
  + breast cancer by measuring the interval (in months) between treatment initiation and disease progression.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1).
Time Frame: At 12 months
Population: Patients on Phase 2 Arm 1 (TP53-mut) - Atezolizumab 840mg IV + Cobimetinib 60mg PO
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2 (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 5
days | 56 [51 to NA] — Could not be estimated from the data due to insufficient number of participants with events

8. Secondary Outcome: Overall Survival (OS) (Phase II) in Days
Description: Assessment of clinical impact (anti-tumor effect) of the combination of atezolizumab and cobimetinib or idasanutiln in patients with metastatic ER
  + breast cancer by measuring the interval (in months) between treatment initiation and death from any cause
Time Frame: At 12 months
Population: Patients on Phase 2 Arm 1 (TP53-mut) - Atezolizumab 840mg IV + Cobimetinib 60mg PO
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2 (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 5
days | 161 [136 to NA] — Could not be estimated from the data due to insufficient number of participants with events.

9. Secondary Outcome: Number of Adverse Events (Phase II)
Description: Assessment of adverse events throughout the phase II study
Time Frame: Up to 28 days after completion of study treatment, for a total of 2 years
Population: patients on atezolizumab and cobimetinib.
Measure: Number; unit: events
Arm/Group | Phase 2 (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 5
events | 99

ADVERSE EVENTS:
Time Frame: Initiation of study medication, throughout the study, and within 28 days (+/- 7 days) of the last dose of study medication, for a total of 2 years.
Arm/Group | Phase 2 (Atezolizumab, Cobimetinib) | Phase 1b - (Atezolizumab, Idasanutlin)
All-Cause Mortality (participants affected / at risk) | 3/5 | 3/7
Serious Adverse Events (participants affected / at risk) | 2/5 | 4/7
Other Adverse Events (participants affected / at risk) | 5/5 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2 (Atezolizumab, Cobimetinib) (N=5) | Phase 1b - (Atezolizumab, Idasanutlin) (N=7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
Suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Strep infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Platelet count decrease (Investigations) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Death (Investigations) | 0 (0) | 1 (1) — Clinical progression
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2 (Atezolizumab, Cobimetinib) (N=5) | Phase 1b - (Atezolizumab, Idasanutlin) (N=7)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 5 (9)
Nausea (Gastrointestinal disorders) | 3 (5) | 5 (12)
Vomiting (Gastrointestinal disorders) | 3 (7) | 4 (7)
Constipation (Gastrointestinal disorders) | 2 (4) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (9)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth ache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (9) | 4 (12)
White blood cell decreased (Investigations) | 3 (8) | 5 (13)
Neutrophil count decreased (Investigations) | 2 (3) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 3 (3)
Platelet count decreased (Investigations) | 1 (2) | 2 (12)
Alanine aminotransferase increased (Investigations) | 3 (6) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2) | 2 (3)
Blood bilirubin increased (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 0 (0) | 1 (1)
GGT increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 4 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5) | 4 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (6) | 2 (2)
Hypokalemia (Investigations) | 3 (5) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (8) | 4 (5)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (6) | 5 (9)
Fever (General disorders) | 1 (2) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (3)
Pain (General disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (5)
Dysgeusia (Nervous system disorders) | 2 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Blurred vison (Eye disorders) | 0 (0) | 2 (2)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT03566485/Prot_SAP_000.pdf